CLINICAL TRIAL: NCT04457219
Title: A Randomised Controlled Trial to Compare Conventional and Haemostatic Dressings to Achieve Rapid and Effective Haemostasis Following Radial Artery Access
Brief Title: Assessment of Radial Artery Complications Whilst Achieving Rapid Haemostasis
Acronym: ARCH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pre-specified interim analysis on data from 2,000 patients by an independent DMSC: recruitment to be stopped early for overwhelming superiority of one of the 3 randomised treatment arms, in the absence of any safety concerns.
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Biolife LLC (Unknown); The Johnson Foundation, United Kingdom (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 271746
Record Dates: First submitted 2020-06-15; First posted 2020-07-07 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Injury; Blood Vessel, Wrist, Radial Artery
Keywords: Rapid; Haemostasis; Hemostasis; Haemostatic; Hemostatic; Statseal; Radial; Comparative Effectiveness Trial; Pragmatic Design; Low-interventional Trial; Transradial; Percutaneous coronary intervention; Coronary angiography
MeSH Terms: conditions — Wounds and Injuries; Fasting

STUDY DESIGN:
Intervention Model Description: 3 arms of randomisation (1:1:1 ratio), parallel treatments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional dressing with 120 minutes external compression (Active Comparator): A standard absorbent dressing is placed on the radial access site, following the transradial angiographic procedure. A radial compression device is then applied to secure patent haemostasis, once the radial sheath is removed. The compression device remains in place for a minimum of 2 hours, as per protocol. This is the standard radial care currently in use at Liverpool Heart and Chest Hospital.
  Interventions: Device: Conventional Dressing; Device: 120 Minutes External Compression
- Conventional dressing with 60 minutes external compression (Experimental): A standard absorbent dressing is placed on the radial access site, following the transradial angiographic procedure. A radial compression device is then applied to secure patent haemostasis, once the radial sheath is removed. The compression device remains in place for a minimum of 1 hour, as per protocol.
  Interventions: Device: Conventional Dressing; Device: 60 Minutes External Compression
- Haemostatic dressing with 60 minutes external compression (Experimental): A haemostatic absorbent dressing is placed on the radial access site, following the transradial angiographic procedure. This consists of a mineral-based dressing that accelerates local haemostasis. A radial compression device is then applied to secure patent haemostasis, once the radial sheath is removed. The compression device remains in place for a minimum of 1 hour, as per protocol.
  Interventions: Device: Haemostatic Dressing; Device: 60 Minutes External Compression

INTERVENTIONS:
Device: Haemostatic Dressing — A Hemostatic Dressing is applied at the radial access site, following a transradial angiographic procedure. This is a mineral-based dressing with a hydrophilic polymer that works independently of the clotting cascade to seal the site, by accelerating topical hemostasis.
  Arms: Haemostatic dressing with 60 minutes external compression
Device: Conventional Dressing — A Conventional Absorbent Dressing is applied at the radial access site, following the transradial angiographic procedure.
  Arms: Conventional dressing with 120 minutes external compression; Conventional dressing with 60 minutes external compression
Device: 120 Minutes External Compression — A radial compression device is applied at the radial access site to achieve patent hemostasis. The device remains in situ for 2 hours. Prolonged time of compression may be required.
  Arms: Conventional dressing with 120 minutes external compression
Device: 60 Minutes External Compression — A radial compression device is applied at the radial access site to achieve patent hemostasis. The device remains in situ for 1 hour. Prolonged time of compression may be required.
  Arms: Conventional dressing with 60 minutes external compression; Haemostatic dressing with 60 minutes external compression

SUMMARY:
The purpose of this study is to compare different protocols aimed at achieving haemostasis (i.e. stop the bleeding) in patients undergoing heart procedures with access through the wrist. Specifically, a haemostatic dressing that aids clotting at the level of the skin will be used and compared with a normal absorbent dressing. Also, a shorter time of compression required to stop the bleeding at the access site will be evaluated.

DETAILED DESCRIPTION:
Radial access for percutaneous cardiac procedures is the preferred method used by most interventional cardiologists. This method has proven to have the least complications and a much quicker patient's recovery time, compared to other access sites (e.g. femoral or brachial). Following sheath removal, a dressing is applied on the skin at the access site. Dressing currently in use include:

1. Conventional absorbent - an absorbent sterile adhesive dressing. This is our current, standard care.
2. Haemostatic - a sterile mineral-based absorbent dressing that aids clotting. It is not currently used at Liverpool Heart and Chest Hospital (LHCH), but it is a licenced product.

A radial compression device is placed over the dressing, and it applies the appropriate amount of mechanical pressure to guarantee patent haemostasis.

This study will recruit patients who are undergoing a cardiac procedure with intended radial access, as part of their standard care. The aim of this study to look at new techniques to reduce the time to successful and complete haemostasis. This may help to expedite patient discharge (avoiding unplanned overnight stay), to reduce nursing times and to decrease the rate of post-procedural, access site-related bleeding and ischemic complications.

At the end of the cardiac procedure, participants will be randomised in a 1:1:1 ratio to one of the following 3 arms:

Arm 1 - conventional absorbent dressing and a compression device applied for 60 mins; Arm 2 - conventional absorbent dressing with a compression device applied for 120 mins (the current standard practice at LHCH); Arm 3 - haemostatic dressing and a compression device applied for 60 mins.

This is a low-interventional, low-risk, pragmatic study comparing strategies that are currently used in every-day clinical practice. The consent seeking process is proportionate and adapted to the design of the study.

Data collection will be electronic and will be performed by medical and nursing staff as part of their normal clinical practice. This will obviate the use of paper-based case record forms.

This study will actively involve medical and nursing staff across the hospital, facilitating multidisciplinary collaboration and integration of clinical research with everyday clinical practice.

ELIGIBILITY:
Pre-Cath Lab Inclusion Criterion:

Patients scheduled for angiographic procedure with proposed radial access, regardless of their gender identity, ethnicity and religious belief

Pre-Cath Lab Exclusion Criteria:

* < 18 years of age
* Planned bilateral radial access
* Any haematoma (> 5 cm in its longest dimension) at planned puncture site prior to radial sheath insertion
* Established diagnosis of any haematologic disorder or genetic defect predisposing to bleeding
* Patients with International Normalised Ratio (INR) > 2.5 prior to the scheduled angiographic procedure
* Inability to perform adequate consent: communication issues (e.g. mental capacity); inadequate time for the participant to read and consider trial; unscheduled Urgent or Emergency procedures i.e. PPCI
* Patients who are scheduled to be transferred to other hospitals ("treat and return") before haemostasis is achieved.
* Electronic Patient Record technical failure leading to an inability to record participants' care

In-Cath Lab Inclusion Criterion:

Single radial sheath in situ with planned removal in lab

In-Cath Lab Exclusion Criteria:

* Sheath removal after 17:00 hrs
* Patient leaving lab with radial sheath in situ
* Trans-ulnar procedure
* Distal (snuffbox) trans-radial procedure
* Any puncture-related haematoma (> 5cm in its longest dimension) prior to radial sheath removal
* Randomisation system not available
* Dressings of both types not available
* A change in patient's clinical condition during procedure deemed by the operator sufficient to exclude from the trial
* Procedural complication requiring procedure termination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2114 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
The rate of failure to achieve haemostasis at the planned compression time | Estimated average of 90 minutes
  After radial sheath is removed and initial haemostasis is secured by Cath Lab team, new overt bleeding or puncture-related haematoma development, occurring out of the Cath Lab, during planned compression period such that:
  * an additional compression device or pressure dressing is applied OR
  * the radial dressing and compression device (either original device or new device) are re-applied de novo OR
  * planned compression duration period to be restarted
  OR
  At the time of planned compression device removal, perceived failure of puncture site haemostasis, manifest as overt bleeding or puncture-related haematoma, that requires re-application of compression (either with the original device, a new device, an additional device, manual compression or a pressure dressing)

SECONDARY OUTCOMES:
Rate of bleeding complications | From randomisation until discharge from hospital, estimated average of 8 hours
  Incidence of bleeding complications related to the arterial puncture. The bleeding complications that will count as secondary outcome measure for the trial will be:
  * Puncture-related haematoma (grades II, III and IV)
  * Vascular surgical or percutaneous intervention for arterial injury or bleeding
Incidence of post-procedural radial artery occlusion | From randomisation until discharge from hospital, estimated average of 8 hours
  Incidence of radial artery occlusion, as a series of parallel, paired comparisons, between the randomised arms of the trial
Time to Haemostasis | From randomisation until discharge from hospital, estimated average of 8 hours
  Time to haemostasis is the interval of time between initial haemostasis following sheath removal and all compression removed, without any compromise in final haemostasis. This outcome measure will report the 'reality' of the time to haemostasis rather than the target period.
Incidence of patients with delayed discharge due to the need for radial access site care | Estimated average 12 hours
  The number and proportion of patients experiencing delayed discharge for reasons related to haemostasis. An analysis plan, including detail of cost-effectiveness model surrounding this outcome, will be produced at a later stage.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney H Stables, Prof, Study Director — Liverpool Heart & Chest Hospital
Locations (1):
- Liverpool Heart & Chest Hospital, Liverpool, Merseyside, United Kingdom